CLINICAL TRIAL: NCT06763107
Title: Validation and Inverse Analysis of The Athletic Shoulder Test (ASH): Reliability of a Novel Upper Body Isometric Strength Test
Brief Title: Validation and Inverse Analysis of The Athletic Shoulder Test (ASH).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Pablo Hernandez-Lucas, Clinical Professor, University of Vigo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DASH
Record Dates: First submitted 2024-12-31; First posted 2025-01-08 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Pain; Sports Physical Therapy
Keywords: Shoulder Pain; Isometric Strength; Muscle Strength Imbalance; Sports Medicine; Rehabilitation
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Validation of isometric shoulder strength tests (ASH and IASH) in high-performance swimmers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Validation of ASH and IASH Tests in Swimmers (Other): Participants perform the Athletic Shoulder (ASH) test and the Inverse Athletic Shoulder (IASH) test to assess isometric shoulder strength at different adduction angles (180º, 135º, 90º) over two sessions. Data is collected to evaluate the reliability and validity of these tests for swimmers.
  Interventions: Procedure: Athletic Shoulder (ASH) and Inverse Athletic Shoulder (IASH) Tests

INTERVENTIONS:
Procedure: Athletic Shoulder (ASH) and Inverse Athletic Shoulder (IASH) Tests — Participants perform the Athletic Shoulder (ASH) test and Inverse Athletic Shoulder (IASH) test to measure maximal isometric shoulder strength in three positions (180º, 135º, 90º) during two separate sessions. Data is used to assess test reliability and validity for high-performance swimmers.

SUMMARY:
To validate both the Athletic Shoulder (ASH) test, conducted on rugby players, and its inverse, the Inverse Athletic Shoulder (IASH) test, for swimmers. This involves assessing the strength relationship between shoulder flexion and extension at three different adduction angles (180º, 135º, 90º) to identify potential injuries associated with these imbalances.

ELIGIBILITY:
Inclusion Criteria:

* High-performance swimmers.
* Aged between 14 and 18 years.
* No acute injuries in the cervical or scapular region.
* Ability to perform the ASH and IASH tests without compensatory movements.

Exclusion Criteria:

* Acute injuries in the cervical or scapular region.
* Inability to maintain proper positioning during the tests due to lack of adequate mobility or strength.
* Refusal to sign informed consent (or legal guardian's consent for minors).

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Intraclass Correlation Coefficient (ICC) for ASH Test | Measured at two time points: baseline (Day 0) and follow-up (Day 2).
  Assessment of between-day reliability of the ASH test using intraclass correlation coefficients (ICC) for shoulder extension at three adduction angles (180º, 135º, 90º).
Intraclass Correlation Coefficient (ICC) for IASH Test | Measured at two time points: baseline (Day 0) and follow-up (Day 2).
  Assessment of between-day reliability of the IASH test using intraclass correlation coefficients (ICC) for shoulder flexion at three adduction angles (180º, 135º, 90º).
Coefficient of Variation (CV) for ASH and IASH Tests | Measured at two time points: baseline (Day 0) and follow-up (Day 2).
  Analysis of the coefficient of variation (CV) to evaluate data dispersion and consistency for both ASH and IASH tests.
Minimum Detectable Change (MDC) for ASH and IASH Tests | Measured at two time points: baseline (Day 0) and follow-up (Day 2).
  Calculation of the minimum detectable change (MDC) to identify the smallest significant change in performance beyond measurement error for both ASH and IASH tests.
Force Ratios Between ASH and IASH Tests | Measured at two time points: baseline (Day 0) and follow-up (Day 2).
  Evaluation of the agonist-antagonist strength ratios between ASH (extension) and IASH (flexion) tests across three adduction angles (180º, 135º, 90º).
Comparison of Shoulder Strength Between Preferred and Non-Preferred Breathing Sides | Measured at two time points: baseline (Day 0) and follow-up (Day 2).
  Analysis of differences in isometric shoulder strength between the preferred and non-preferred breathing sides in ASH and IASH tests across three adduction angles.
Evaluation of Test Fatigue and Its Impact on Reliability | Measured at two time points: baseline (Day 0) and follow-up (Day 2).
  Assessment of fatigue effects during ASH and IASH tests, considering the 20-second rest period and total number of efforts (36 per participant), and their potential impact on test reliability and strength measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Pablo, Pontevedra, Spain